CLINICAL TRIAL: NCT01525797
Title: Immunomonitoring of Transplant Patients
Brief Title: Blood Draw Study for Liver Transplant Patients
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 002-197
Record Dates: First submitted 2011-05-11; First posted 2012-02-03 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Liver Transplant Recipients
Keywords: Liver Transplant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control
- Rejection

SUMMARY:
The purpose of this study is to see what a lab test will show and if there is a way to predict which patients will be more likely to have rejection after receiving a liver transplant.

DETAILED DESCRIPTION:
The purpose of this study is simply to see what the new oligonucleotide microarrays will show when comparing the the different patient groups. The results of this study will be one of the first steps In exploring the potential use of this new test.

ELIGIBILITY:
Inclusion Criteria:

* Received a liver Transplant

Exclusion Criteria:

* Received Multiple Organ Transplant

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Liver Clinic
Sampling Method: Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2002-10-15 (Actual); Primary Completion 2013-10-04 (Actual); Study Completion 2013-10-04 (Actual)

PRIMARY OUTCOMES:
Identify signatures predictive of graft rejection or tolerance. | 2 years
  Analyze the pattern of gene expression in patients undergoing solid organ transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Goran Klintmalm, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States